CLINICAL TRIAL: NCT05528146
Title: Effects of Psyllium on Constipation in Schizophrenic: A Randomized Controlled Crossover Trial
Brief Title: Effects of Psyllium on Constipation in Schizo-phrenic: A Randomized Controlled Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Wang Chin Hsiu, Nurse Practitioner, Hungkuang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Hungkuang University
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia; Constipation
Keywords: Schizophrenia; Psyllium; Constipation
MeSH Terms: conditions — Schizophrenia; Constipation

STUDY DESIGN:
Intervention Model Description: During the first stage, both groups underwent pre-tests before the intervention. In the second stage, the two groups separately received a daily intake of 3.5 grams and 7 grams of psyllium husk for four weeks, followed by the first post-test. There was then a one-week washout period. In the third stage, the two groups switched the intake dosage of psyllium husk and underwent the second post-test after another four weeks of continuous intake.
Who Masked: Participant
Masking Description: The study employed a single-blind and simple randomization approach, with hospital wards divided into two groups. Only Researchers Know Psyllium Dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group for women (Experimental): In a single-blind crossover trial (male or female), these groups will receive 3.5 g/day or 7 g/day of psyllium for 4 weeks. The trial will stop 1 week after the first phase and post-test. The two groups will then swap doses for 4 weeks. Post-tests will be recorded upon completion of this Phase 2 trial. After completing the trial, determine the dose effect.
  Interventions: Dietary Supplement: Psyllium huks
- B group for man (Experimental): In a single-blind crossover trial (male or female), these groups will receive 3.5 g/day or 7 g/day of psyllium for 4 weeks. The trial will stop 1 week after the first phase and post-test. The two groups will then swap doses for 4 weeks. Post-tests will be recorded upon completion of this Phase 2 trial. After completing the trial, determine the dose effect.
  Interventions: Dietary Supplement: Psyllium huks

INTERVENTIONS:
Dietary Supplement: Psyllium huks — psyllium in 250ml of water

SUMMARY:
Constipation in schizophrenia is an important issue in clinical care. Constipation needs psychiatric professionals concerning and providing intervention because it may cause ileus and lead to death. The cause of constipation in patients may be due to side effects of antipsychotic medication, sedentary lifestyle, insufficient water intake, fiber, etc. The study aims to increase fiber of the consumption of psyllium to assess the constipation effectiveness in schizophrenics. The study conducted a crossover research design. G-power was used to calculate the 22 subjects in each of the two groups. A total of 44 patients with constipation who were schizophrenics will participate in the study. Patients will use simple randomly to be divided into two groups based on their live ward for pre-testing. These two groups will receive either psyllium 3.5 g/day or 7 g/day for 4 weeks in a single-blind, crossover trial. The trial will stop 1week after the first phase and post-test. Then, two groups will exchange the dose for 4 weeks. Post-test will record after finishing this second phase trial. This study can understand the benefits of psyllium on schizophrenics with constipation symptoms and can give professional suggestions to patients with constipation in the future.

DETAILED DESCRIPTION:
The study was conducted in the psychiatric department of a hospital in the central region and utilized a crossover design involving a total of 42 patients with schizophrenia. The study employed a single-blind and simple randomization approach, with hospital wards divided into two groups. During the first stage, both groups underwent pre-tests before the intervention. In the second stage, the two groups separately received a daily intake of 3.5 grams and 7 grams of psyllium husk for four weeks, followed by the first post-test. There was then a one-week washout period. In the third stage, the two groups switched the intake dosage of psyllium husk and underwent the second post-test after another four weeks of continuous intake. The research findings showed significant improvements in the frequency of constipation, stool consistency, and subjective experience of bowel movements in patients with schizophrenia following the intervention with psyllium husk.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-V was diagnoses with schizophrenia inpatients.
2. Aged between 20 years and above.
3. Those who defecate less than 3 times a week, or those who have Bristol stool form scale between 1 and 2, or those who have constipation assessment scale (CAS) scores more than one point from questions 3 to 8; Or use PRN stool softeners (including oral and suppository) at least once a week.
4. Clear awareness and able to communicate in Chinese and Taiwanese.

Exclusion Criteria:

1. Patients with intestinal diseases such as colon cancer, irritable bowel syndrome and other organic intestinal diseases such as rectal bleeding, intestinal surgery, rectal prolapse and other medical history.
2. Cases with positive fecal occult blood test in the past six months, changes in stool thickness for one month, history of iron deficiency anemia, and unexplained weight loss for one month.
3. Those who are unable to cooperate due to obvious mental symptoms.
4. History of grain allergy, asthma.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
frequency of constipation | 4weeks
  To assess the outcome measure of constipation frequency, researchers will collect the number of weekly bowel movements from participants by daily inquiries. Constipation, in this context, is defined as having fewer than three bowel movements per week. Additionally, researchers will record any associated discomfort or symptoms related to constipation.
  Wilcoxon Signed Rank Test analysis showed a significant difference between the pre-test and the second stage (3.5 g/day psyllium) (z = -2.08, p = .04), Cohen's d = .39; the pre-test and the three stage (7 g/day psyllium), there was a statistically significant difference (z = -2.2, p = .03) , Cohen's d = .42

SECONDARY OUTCOMES:
Stool type(bristol stool form) | 4weeks
  To assess the outcome measure of stool consistency, researchers will utilize the Bristol Stool Scale, which categorizes stool types into seven categories. These categories will be further classified into three groups: constipation, normal, and diarrhea. Constipation, in this context, is defined as the presence of stool types falling within the constipation category, as specified on the Bristol Stool Scale. Researchers will collect this data through daily inquiries with participants and record any associated discomfort or symptoms related to constipation.
  The Wilcoxon Signed Rank Test counted the stool patterns of the subjects and found that when taking 3.5g/day psyllium husk, the constipation pattern was reduced (z = -3.08, p = .002, Cohen's d= .54) , the amount of effect was reached; and the normal stool pattern increased (z = -4.35, p = < .001, Cohen's d = - .89).

OTHER OUTCOMES:
Constipation Assessment Scale, CAS | 4weeks
  After the completion of the four-week study period, researchers will conduct a Constipation Assessment Scale (CAS) assessment to evaluate participants' perception of constipation. A higher CAS score indicates more severe constipation symptoms. Additionally, researchers will inquire with participants every four weeks to collect data on their perception of constipation and record any associated discomfort or symptoms.
  The Wilcoxon Signed Rank Test compared the intake of 3.5 g/day psyllium husk before the pre-test, and the subjective feeling of constipation with 3.5 g/day psyllium husk decreased significantly, reaching a statistical difference (z = -3.94, p = <.001), Cohen's d = 1.08,

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Hospitol, Chang-hua, Puxin Township, Taiwan

IPD SHARING:
Plan to Share IPD: No